CLINICAL TRIAL: NCT02726009
Title: An Open-label, Single-Arm, Multicenter, Phase IV Trial to Evaluate the Safety of Firmagon® in Androgen Deprivation Therapy in Indian Patients Diagnosed With Advanced Hormone-dependent Prostate Cancer
Brief Title: A Trial to Evaluate Safety of Firmagon® (Degarelix) in Indian Patients Diagnosed With Advanced Hormone-dependent Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000201
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix (Experimental)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix
  Other Names: Firmagon®

SUMMARY:
The purpose of this open-label, single-arm, multicenter, post-marketing trial is to evaluate long-term safety of Firmagon® in approximately 230 Indian patients diagnosed with advanced hormone-dependent prostate cancer requiring androgen deprivation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent before any study-related activity is performed
* Advanced hormone-dependent prostate cancer for which androgen deprivation therapy is indicated, and independently from this trial, Firmagon® is intended to be used for treatment
* Age greater than or equal to 18 years and less than 80 years
* Advanced hormone-dependent prostate cancer without any other clinically significant disorder
* Easten Cooperative Oncology Group score ≤ 2
* PSA ≥ 2 ng/mL at screening
* Life expectancy of at least 12 months as per the investigator's judgement

Exclusion Criteria:

* Previous or concurrent hormonal management of prostate cancer
* Contraindication for prescription of Firmagon®
* Concurrent treatment with a 5-α-reductase inhibitor
* Considered as a candidate for curative therapy
* History of severe untreated asthma, anaphylactic reactions or severe urticaria and/or angioedema
* QTc interval over 450 msec or risk factors for torsades de pointes or on Class IA and Class III anti arrhythmic medications
* Cancer within the last 5 years except prostate cancer and surgically removed basal or squamous cell carcinoma of the skin
* Known or suspected hepatic, symptomatic biliary disease (this includes moderate to severe chronic hepatic impairment)
* Patients with clinically significant laboratory abnormalities / disorders other than prostate cancer
* Patient with Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) infections

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | Up to Day 364
Severity of adverse events | Up to Day 364
Clinically significant changes in laboratory values (hematology and clinical biochemistry) | From baseline to Day 364
Clinically significant changes in vital signs | From baseline to Day 364

SECONDARY OUTCOMES:
Cumulative probability of no Prostate Specific Antigen (PSA) failure | Up to Day 364
  PSA failure defined as an increase in serum PSA of 50%, and at least 5 ng/mL, compared to nadir, measured on two consecutive occasions at least 2 weeks apart
Cumulative probability of Progression Free Survival (PFS) | Up to Day 364
  PFS defined as PSA failure, death from any cause, or introduction of additional therapy related to prostate cancer, whichever is first
Change in International Prostate Symptom Score (IPSS) | From baseline to Day 364
Change in physician's satisfaction score | From baseline to Day 364

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (19):
- India (19):
  - S. P Medical College and AG of Hospitals, Bikaner, Rajasthan
  - Krishna Institute of Medical Sciences, Secunderabad, Telangana
  - Bodyline Hospitals, Ahmedabad
  - HCG Multi Specialty Hospital, Ahmedabad
  - Shalby Hospital, Ahmedabad
  - HealthCare Global Enterprises Limited, Bangalore
  - KLE's Dr. Prabhakar Kore Hospital & MRC, Belagavi
  - Apollo Speciality Hospital, Chennai
  - Rajiv Gandhi Cancer Institute and Research Centre, Delhi
  - Muljibhai Patel Urological Hospital, Gujrāt
  - CHL Hospital, Indore
  - SMS Medical College & Attached Hospital's, Jaipur
  - Tata Medical Center, Kolkata
  - King's George Medical University, Lucknow
  - Kokilaben Dhirubhai Ambani Hospital and Medical Research Institute, Mumbai
  - Tata Memorial Hospital, Mumbai
  - Government Medical College and Super Specialty Hospital, Nagpur
  - Rml & Pgimer, New Delhi
  - Aman Hospital and Research Center, Vadodara